CLINICAL TRIAL: NCT03637569
Title: The Relationship Between Triceps Skinfold and Overall Survival of Pancreatic Cancer, Cholangiocarcinoma and Gallbladder Cancer.
Brief Title: The Relationship Between Triceps Skinfold and Overall Survival of Pancreas, Bile Duct, Gallbladder Cancer
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JooKyung Park, Assistant Professor, Samsung Medical Center
Other Study IDs: SMC 2018-04-087-001
Record Dates: First submitted 2018-07-26; First posted 2018-08-20 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Pancreas Cancer; Cholangiocarcinoma; Gallbladder Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients: Newly diagnosed pancreatic, bile duct or GB cancer patients at samsung medical center.
  Interventions: Other: Measurement of triceps skinfold thickness

INTERVENTIONS:
Other: Measurement of triceps skinfold thickness — By using skin thickness caliper, measure triceps skinfold thickness on the half of forearm (Rt side). In every 3 weeks, triceps skinfold thickness will be measured.

SUMMARY:
In this study, the investigators aim to demonstration of relationship between triceps skinfold thickness and overall survival of pancreatic cancer, cholangiocarcinoma and GB cancer.

DETAILED DESCRIPTION:
Cachexia is frequently seen in pancreatic cancer(70-80%) and associated with reduced survival, reduced treatment tolerance and reduction in QoL. In recent studies, low-normal BMI have worse outcome (overall mortality) in cardiovascular, malignant, chronic disease (So called "obesity paradox") BMI is simple method but hard to define body composition because BMI is based on only weight and height. Skinfold thickness is strongly associated with body fatness than BMI. In this study, the ivestigators aim to demonstration of relationship between triceps skinfold thickness and overall survival of pancreatic cancer, cholangiocarcinoma and GB cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed pancreatic, bile duct or gallbladder cancer patients, undergoing therapeutic management (including surgery, chemotherapy or palliative care).
* Age above 18 years old

Exclusion Criteria:

* Other malignant disease
* Underlying intestinal disease that cause absorprtion disorder
* Underlying psychiatric disorder such as eating disorder (bulimia, anorexia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visit and treated at Samsung medical center.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | through study completion, an average of 2 year
  The duration between diagnosis and death

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No